CLINICAL TRIAL: NCT04765033
Title: Efficacy of Nebulised 5% Hypertonic Saline in Children With Chronic Suppurative Lung Disease
Brief Title: Trial on The Efficacy of Hypertonic Saline on Non-CF CSLD.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Anna Marie Nathan, Consultant and Professor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020729-8926
Record Dates: First submitted 2021-02-08; First posted 2021-02-21 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Bronchiectasis
Keywords: CSLD; Child; Nebuliser; Hypertonic Saline; Outcome; Chronic cough
MeSH Terms: conditions — Bronchiectasis; Chronic Cough | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: Double-blind Placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5% Hypertonic saline (Active Comparator): 5% hypertonic saline nebuliser 4 mls twice in a day for 3 months
  Interventions: Drug: Nebulized 5% Hypertonic saline
- Placebo (Placebo Comparator): 0.9% saline nebuliser 4 mls twice in a day for 3 months
  Interventions: Drug: Nebulized 5% Hypertonic saline

INTERVENTIONS:
Drug: Nebulized 5% Hypertonic saline — nebulized 0.9% saline
  Other Names: Placebo

SUMMARY:
To determine the efficacy of nebulized 5% hypertonic saline on cough severity and quality of life, in children with non-CF CSLD.

Secondary Aims:

To determine the:

1. Efficacy of nebulized 5% hypertonic saline on airway microbiome, pulmonary exacerbation rate, healthcare utilization, and rescue antibiotics.
2. Efficacy of nebulized 5% hypertonic saline on lung function
3. Adverse effects of nebulized 5% hypertonic saline in children

DETAILED DESCRIPTION:
Primary Aim:

To determine the efficacy of nebulized 5% hypertonic saline on cough severity and quality of life, in children with non-CF CSLD.

Here the investigators will be using validated pediatric cough questionnaires to asses this. Patients will answer these questionnaires at first recruitment ( -1 mth), at randomization (0 month) and after 3 mths of use of the nebulized study drug (+ 3 mths)

Secondary Aims:

To determine the:

1. Efficacy of nebulized 5% hypertonic saline on the airway microbiome, pulmonary exacerbation rate, healthcare utilization, and rescue antibiotics.

   Here the investigators will be taking history on the exacerbations, use of antibiotics and healthcare utilization before and after use of the hypertonic saline. Furthermore, Nasopharyngeal swabs will be done to review possible changes in microbiota, again before and after use of the 5% HS.
2. Efficacy of nebulized 5% hypertonic saline on lung function. Here is investigators will be doing portable spirometry ( pre and post bronchodilator).

   Patients will perform at randomization (0 month) and after 3 mths of use of the nebulized study drug (+ 3 mths)
3. Adverse effects of nebulized 5% hypertonic saline in children HS has been associated with side-effects. The investigators will monitor this. We will asses presence of these symptoms at randomization (0 month) and after 3 mths of use of the nebulized study drug (+ 3 mths) to ensure these are from the nebulizer.

ELIGIBILITY:
Inclusion Criteria:

* Patients < 18 years old
* Followed up in the paediatric respiratory clinic of UMMC with a diagnosis of CSLD

Exclusion Criteria:

* Incomplete data or refusal to participate
* Unwell and/or unable to stop HS and/or antibiotics of any preparation other than azithromycin ( EOD
* On supplementary oxygen/home ventilation
* Poorly controlled asthma (as in the GINA guidelines) or bronchoconstriction that precedes the use of hypertonic saline.
* Oral antibiotics for less than 4 weeks before randomization for medication.
* Fall in PEFR > 20% post 5% HS challenge test or a positive HS challenge test in young children, as mentioned below.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Change in the Short Parent-proxy cough quality of life (PC-QOL) score | at -1 month of randomization, at day 1 of randomization, at 3 months of use of study drug
  Short PCQOL: This is a validated cough quality-of-life(QoL) questionnaire for parents of children with chronic cough, with a translated Malay version. Minimal Important Difference(MID) of 0.9 has been found in the validation study.
  The answers are on a Likert scale from 1 (every time) to 7( none). A lower score denotes a lower quality of life.
  The patients will answer either the English or the translated Malay version
Change in the Chronic Cough-specific QoL(CC-QOL) score | at -1 month of randomization, at day 1 of randomization, at 3 months of use of study drug
  Chronic cough-specific QOL: This is a validated cough QoL questionnaire to be answered by children 7 years till 18 years old with a MID of about 1.1. The answers are in a Likert scale from 1 ( every time) to 7( none). A lower score denotes a lower quality of life.
  The patients will answer either the English or the translated Malay version

SECONDARY OUTCOMES:
Airway microbiome | At day 1 of randomization, at 3 months of use of study drug
  DNA will be extracted from swabs using the Qiagen DNA Isolation Kit in accordance with the manufacturer's instructions. Bacterial profiling utilised the 16S rRNA gene targeting variable regions V3 - V4 will be carried out using Nextseq 2500 platform. Resulting raw fastq data will be processed using Dada2 R package and exported into phyloseq Rprogram for downstream analysis. The Alpha diversity will be measured using the Shannon and Simpson diversity indices while the beta diversity will be accessed using principle coordinate analysis and Permutational multivariate analysis of variance(PERMANOVA). Differentially abundant taxa will be identified by comparing the fold-change different using DESeq2.
Number of Exacerbations | at -1 month of randomization, at day 1 of randomization, at 3 months of use of study drug
  Defined as having one major and 2 minor OR 2 major criteria irrespective of whether antibiotics are prescribed.
  Criteria for exacerbation:
  Major: (1) Wet cough over 72 hours, (2) Severe cough over 72 hours Minor: (1) Change in Sputum colour, (2) Chest pain, (3) SOB, (4) Haemoptysis, (5) + ve Chest signs
  At -1 month, we will look at the no of exacerbations in the past 1 year. Before the use of the study drug and after 3 months of use of the study drug, we will look at the no of exacerbations in the preceding 1 month and 3 months, respectively.
Number of Unscheduled Health Care Visits | at -1 month of randomization, at day 1 of randomization, at 3 months of use of study drug
  any unscheduled doctor visits for cough, shortness of breath or any other respiratory associated symptom.
  This will be for the last 3 months before day 1 of randomization and after 3 months of use of study drug
No of episodes of rescue antibiotics | at -1 month of randomization, at day 1 of randomization, at 3 months of use of study drug
  Prescription of antibiotics (including nebulized antibiotics) at least for 3 days for respiratory associated symptoms.
  This will be in the past 3 months, before randomization and during the next 3 months, while on the study drug.
FEV1 | At day 1 of randomization, at 3 months of use of study drug
  FEV1 will be performed in sitting position(both pre and post 4 puffs of MDI Salbutamol) using the portable spirometry, performed in clinic. The best spirometric measure of at least 3 reproducible attempts will be recorded for analysis. Reference values from Morris/Polgar will be used with ethnic corrections. FEV1 value will be converted into z-score by using GrowingLungs software.
FVC | At day 1 of randomization, at 3 months of use of study drug
  FVC will be performed in sitting position(both pre and post 4 puffs of MDI Salbutamol) using the portable spirometry, performed in clinic. The best spirometric measure of at least 3 reproducible attempts will be recorded for analysis. Reference values from Morris/Polgar will be used with ethnic corrections. FVC value will be converted into z-score by using GrowingLungs software.
FEF 25-75% | At day 1 of randomization, at 3 months of use of study drug
  FEF 25-75% will be performed in sitting position(both pre and post 4 puffs of MDI Salbutamol) using the portable spirometry, performed in clinic. The best spirometric measure of at least 3 reproducible attempts will be recorded for analysis. Reference values from Morris/Polgar will be used with ethnic corrections. FEF25-75% value will be converted into z-score by using GrowingLungs software.
PEFR ( pre and post), if possible | at -1 month of randomization, at day 1 of randomization, at 3 months of use of study drug
  The best PEFR measure out of 3 reproducible attempts ( both pre and post 4 puffs of MDI Salbutamol), performed when relatively well and stable, will be recorded for analysis.
Cough diary | at -1 month of randomization, at day 1 of randomization, at 3 months of use of study drug
  The cough score will be assessed using the Malay version, used in the HOspitalised Pneumonia Extended study, whereby the cough score will be tabulated daily.
  The cough diary has recordings for both day time cough: score 0 ( no cough) till score 5 ( Cannot perform most usual day-time activity due to severe coughing).
  The night cough is scored score 0 ( no cough) till score 5 ( distressing cough.).
  A higher score indicates more severe cough.
Number of Adverse events | At day 1 of randomization, at 3 months of use of study drug
  cough, haemoptysis, sore throat, throat burning, chest tightness, hoarseness of voice.

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Nathan, Principal Investigator — UMMC
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Lembah Pantai, Malaysia

IPD SHARING:
Plan to Share IPD: No
Not to share

REFERENCES:
- [Result] McCallum GB, Binks MJ. The Epidemiology of Chronic Suppurative Lung Disease and Bronchiectasis in Children and Adolescents. Front Pediatr. 2017 Feb 20;5:27. doi: 10.3389/fped.2017.00027. eCollection 2017. PMID 28265556
- [Result] Lovie-Toon YG, Grimwood K, Byrnes CA, Goyal V, Busch G, Masters IB, Marchant JM, Buntain H, O'Grady KF, Chang AB. Health-resource use and quality of life in children with bronchiectasis: a multi-center pilot cohort study. BMC Health Serv Res. 2019 Aug 13;19(1):561. doi: 10.1186/s12913-019-4414-5. PMID 31409413
- [Result] Chang AB, Bush A, Grimwood K. Bronchiectasis in children: diagnosis and treatment. Lancet. 2018 Sep 8;392(10150):866-879. doi: 10.1016/S0140-6736(18)31554-X. PMID 30215382
- [Result] Nathan AM, Muthusamy A, Thavagnanam S, Hashim A, de Bruyne J. Chronic suppurative lung disease in a developing country: impact on child and parent. Pediatr Pulmonol. 2014 May;49(5):435-40. doi: 10.1002/ppul.23001. Epub 2014 Jan 31. PMID 24482322
- [Result] Kumar A, Lodha R, Kumar P, Kabra SK. Non-cystic fibrosis bronchiectasis in children: clinical profile, etiology and outcome. Indian Pediatr. 2015 Jan;52(1):35-7. doi: 10.1007/s13312-015-0563-8. PMID 25638182
- [Result] Kapur N, Masters IB, Newcombe P, Chang AB. The burden of disease in pediatric non-cystic fibrosis bronchiectasis. Chest. 2012 Apr;141(4):1018-1024. doi: 10.1378/chest.11-0679. Epub 2011 Sep 1. PMID 21885727
- [Result] Gaillard EA, Carty H, Heaf D, Smyth RL. Reversible bronchial dilatation in children: comparison of serial high-resolution computer tomography scans of the lungs. Eur J Radiol. 2003 Sep;47(3):215-20. doi: 10.1016/s0720-048x(02)00122-5. PMID 12927665
- [Result] Cole PJ. Inflammation: a two-edged sword--the model of bronchiectasis. Eur J Respir Dis Suppl. 1986;147:6-15. PMID 3533593
- [Result] Hahn A, Warnken S, Perez-Losada M, Freishtat RJ, Crandall KA. Microbial diversity within the airway microbiome in chronic pediatric lung diseases. Infect Genet Evol. 2018 Sep;63:316-325. doi: 10.1016/j.meegid.2017.12.006. Epub 2017 Dec 7. PMID 29225146
- [Result] Zemanick ET, Harris JK, Wagner BD, Robertson CE, Sagel SD, Stevens MJ, Accurso FJ, Laguna TA. Inflammation and airway microbiota during cystic fibrosis pulmonary exacerbations. PLoS One. 2013 Apr 30;8(4):e62917. doi: 10.1371/journal.pone.0062917. Print 2013. PMID 23646159
- [Result] Cox MJ, Allgaier M, Taylor B, Baek MS, Huang YJ, Daly RA, Karaoz U, Andersen GL, Brown R, Fujimura KE, Wu B, Tran D, Koff J, Kleinhenz ME, Nielson D, Brodie EL, Lynch SV. Airway microbiota and pathogen abundance in age-stratified cystic fibrosis patients. PLoS One. 2010 Jun 23;5(6):e11044. doi: 10.1371/journal.pone.0011044. PMID 20585638
- [Result] Prentice BJ, Wales S, Doumit M, Owens L, Widger J. Children with bronchiectasis have poorer lung function than those with cystic fibrosis and do not receive the same standard of care. Pediatr Pulmonol. 2019 Dec;54(12):1921-1926. doi: 10.1002/ppul.24491. Epub 2019 Sep 1. PMID 31475469
- [Result] Chang AB. Bronchiectasis: so much yet to learn and to do. Paediatr Respir Rev. 2011 Jun;12(2):89-90. doi: 10.1016/j.prrv.2011.01.001. Epub 2011 Feb 2. No abstract available. PMID 21458735
- [Result] Tarran R, Grubb BR, Parsons D, Picher M, Hirsh AJ, Davis CW, Boucher RC. The CF salt controversy: in vivo observations and therapeutic approaches. Mol Cell. 2001 Jul;8(1):149-58. doi: 10.1016/s1097-2765(01)00286-6. PMID 11511368
- [Result] Kerem E, Reisman J, Corey M, Canny GJ, Levison H. Prediction of mortality in patients with cystic fibrosis. N Engl J Med. 1992 Apr 30;326(18):1187-91. doi: 10.1056/NEJM199204303261804. PMID 1285737
- [Result] Reeves EP, Williamson M, O'Neill SJ, Greally P, McElvaney NG. Nebulized hypertonic saline decreases IL-8 in sputum of patients with cystic fibrosis. Am J Respir Crit Care Med. 2011 Jun 1;183(11):1517-23. doi: 10.1164/rccm.201101-0072OC. Epub 2011 Feb 17. PMID 21330456
- [Result] Elkins MR, Bye PT. Inhaled hypertonic saline as a therapy for cystic fibrosis. Curr Opin Pulm Med. 2006 Nov;12(6):445-52. doi: 10.1097/01.mcp.0000245714.89632.b2. PMID 17053496
- [Result] Dellon EP, Donaldson SH, Johnson R, Davis SD. Safety and tolerability of inhaled hypertonic saline in young children with cystic fibrosis. Pediatr Pulmonol. 2008 Nov;43(11):1100-1106. doi: 10.1002/ppul.20909. PMID 18828160
- [Result] Kellett F, Redfern J, Niven RM. Evaluation of nebulised hypertonic saline (7%) as an adjunct to physiotherapy in patients with stable bronchiectasis. Respir Med. 2005 Jan;99(1):27-31. doi: 10.1016/j.rmed.2004.05.006. PMID 15672845
- [Result] Kellett F, Robert NM. Nebulised 7% hypertonic saline improves lung function and quality of life in bronchiectasis. Respir Med. 2011 Dec;105(12):1831-5. doi: 10.1016/j.rmed.2011.07.019. Epub 2011 Oct 22. PMID 22018993
- [Result] Nicolson CH, Stirling RG, Borg BM, Button BM, Wilson JW, Holland AE. The long term effect of inhaled hypertonic saline 6% in non-cystic fibrosis bronchiectasis. Respir Med. 2012 May;106(5):661-7. doi: 10.1016/j.rmed.2011.12.021. Epub 2012 Feb 19. PMID 22349069
- [Result] Paff T, Daniels JM, Weersink EJ, Lutter R, Vonk Noordegraaf A, Haarman EG. A randomised controlled trial on the effect of inhaled hypertonic saline on quality of life in primary ciliary dyskinesia. Eur Respir J. 2017 Feb 23;49(2):1601770. doi: 10.1183/13993003.01770-2016. Print 2017 Feb. PMID 28232410
- [Result] Sidhu MK, Mandal P, Hill AT. Developing drug therapies in bronchiectasis. Expert Opin Investig Drugs. 2015 Feb;24(2):169-81. doi: 10.1517/13543784.2015.971153. Epub 2014 Oct 11. PMID 25307313
- [Result] Goyal V, Grimwood K, Marchant J, Masters IB, Chang AB. Does failed chronic wet cough response to antibiotics predict bronchiectasis? Arch Dis Child. 2014 Jun;99(6):522-5. doi: 10.1136/archdischild-2013-304793. Epub 2014 Feb 12. PMID 24521788
- [Result] Chang AB, Boyce NC, Masters IB, Torzillo PJ, Masel JP. Bronchoscopic findings in children with non-cystic fibrosis chronic suppurative lung disease. Thorax. 2002 Nov;57(11):935-8. doi: 10.1136/thorax.57.11.935. PMID 12403874
- [Result] Kapur N, Masel JP, Watson D, Masters IB, Chang AB. Bronchoarterial ratio on high-resolution CT scan of the chest in children without pulmonary pathology: need to redefine bronchial dilatation. Chest. 2011 Jun;139(6):1445-1450. doi: 10.1378/chest.10-1763. Epub 2010 Sep 23. PMID 20864608
- [Result] Newcombe PA, Sheffield JK, Petsky HL, Marchant JM, Willis C, Chang AB. A child chronic cough-specific quality of life measure: development and validation. Thorax. 2016 Aug;71(8):695-700. doi: 10.1136/thoraxjnl-2015-207473. Epub 2016 Feb 3. PMID 26842959
- [Result] Callahan BJ, McMurdie PJ, Rosen MJ, Han AW, Johnson AJ, Holmes SP. DADA2: High-resolution sample inference from Illumina amplicon data. Nat Methods. 2016 Jul;13(7):581-3. doi: 10.1038/nmeth.3869. Epub 2016 May 23. PMID 27214047
- [Result] McMurdie PJ, Holmes S. phyloseq: an R package for reproducible interactive analysis and graphics of microbiome census data. PLoS One. 2013 Apr 22;8(4):e61217. doi: 10.1371/journal.pone.0061217. Print 2013. PMID 23630581
- [Result] Love MI, Huber W, Anders S. Moderated estimation of fold change and dispersion for RNA-seq data with DESeq2. Genome Biol. 2014;15(12):550. doi: 10.1186/s13059-014-0550-8. PMID 25516281
- [Result] Chang AB, Fong SM, Yeo TW, Ware RS, McCallum GB, Nathan AM, Ooi MH, de Bruyne J, Byrnes CA, Lee B, Nachiappan N, Saari N, Torzillo P, Smith-Vaughan H, Morris PS, Upham JW, Grimwood K. HOspitalised Pneumonia Extended (HOPE) Study to reduce the long-term effects of childhood pneumonia: protocol for a multicentre, double-blind, parallel, superiority randomised controlled trial. BMJ Open. 2019 Apr 24;9(4):e026411. doi: 10.1136/bmjopen-2018-026411. PMID 31023759
- [Result] Kapur N, Masters IB, Morris PS, Galligan J, Ware R, Chang AB. Defining pulmonary exacerbation in children with non-cystic fibrosis bronchiectasis. Pediatr Pulmonol. 2012 Jan;47(1):68-75. doi: 10.1002/ppul.21518. Epub 2011 Aug 9. PMID 21830316
- [Result] Stanojevic S, Wade A, Stocks J, Hankinson J, Coates AL, Pan H, Rosenthal M, Corey M, Lebecque P, Cole TJ. Reference ranges for spirometry across all ages: a new approach. Am J Respir Crit Care Med. 2008 Feb 1;177(3):253-60. doi: 10.1164/rccm.200708-1248OC. Epub 2007 Nov 15. PMID 18006882
- [Result] Walker PP, Key AL. How to perform peak flow and spirometry tests. BMJ. 2016 May 11;353:h6159. doi: 10.1136/sbmj.h6159. No abstract available. PMID 31055386
- [Result] Newcombe PA, Sheffield JK, Chang AB. Parent cough-specific quality of life: development and validation of a short form. J Allergy Clin Immunol. 2013 Apr;131(4):1069-74. doi: 10.1016/j.jaci.2012.10.004. Epub 2012 Nov 10. PMID 23146374